CLINICAL TRIAL: NCT05650645
Title: The Efficacy of Incobotulinum Toxin A Injections for Treatment of Tinnitus: a Randomized Controlled Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PMR-2021-29462
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Incobotulinium toxin A group (Experimental): Individuals with symptoms of tetanus will receive three serial injections of incobotulinum toxin A into the auricular muscles.
  Interventions: Drug: incobotulinum toxin A
- Placebo (Placebo Comparator): Individuals with symptoms of tetanus will receive placebo saline injections.
  Interventions: Drug: Placebo-Saline

INTERVENTIONS:
Drug: incobotulinum toxin A — The study intervention is a syringe of 50 units of incobotulinum toxin A total, with 25 units per side, a total of 6 injection sites incobotulinum toxin A diluted into 1 ml of normal saline, injected in equal amounts into the anterior, superior, and posterior auricular muscles using anatomical landmarks. This will be approximately 0.16 mL (8-9 units) of the combined solution per injection site.
  Arms: Incobotulinium toxin A group
Drug: Placebo-Saline — Placebo injections will be preservative free normal saline. Injections will be administered similar to the drug injections.
  Arms: Placebo

SUMMARY:
Tinnitus is a persistent non-physiologic, non-psychiatric, ringing in the ear that affects up to 20% of the general US population. The purpose of this study is to assess the patient reported effectiveness of Xeomin (incobotulinumtoxinA) injections into the auricular muscles for relief of tinnitus with use of the Tinnitus Handicap Inventory questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 or older
* Unilateral or bilateral tinnitus present for ≥ 2 months
* A score >16 on the Tinnitus Handicap Inventory
* Participants must be willing and able to provide informed consent.

Exclusion Criteria:

* Patients with known hypersensitivity to any botulinum toxin product or to any of the components in the formulation.
* Patients who have received botulinum toxin injections for any medical reason within 4 months prior to screening.
* Patients with infection at proposed injection sites.
* Patients scheduled for neurological or otological surgery for chronic ear disease, vestibular schwannoma, meningioma, or skull base tumors.
* Significant psychiatric history or associated diagnosis of major depression.
* Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-29 (Actual); Study Completion 2025-12-29 (Actual)

PRIMARY OUTCOMES:
Change in the Tinnitus Handicap Inventory score | pre-injection baseline to 4-6 weeks post injection
  in the group assigned to placebo for the first stage

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Standal, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States